CLINICAL TRIAL: NCT07163468
Title: Neuromusculoskeletal Alterations After ACL Injury: A Cross-Sectional Study of Cortical Activity, Motor Response, and Psychological Readiness
Brief Title: Neuromusculoskeletal Alterations After ACL Injury
Acronym: NEURO-ACL
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Veysel Uludag, Lecturer, Duzce University
Other Study IDs: 2025/177
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Injuries; Sports Injury; Neurocognitive Function
Keywords: Anterior Cruciate Ligament; Kinesiophobia; Electroencephalography
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Athletic Injuries; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Control Group: Athletes with no history of knee injury or surgery (n=20).
- Primary ACL Reconstruction Group: Athletes who had undergone a single ACL reconstruction, with rehabilitation completed at least 6 months prior to enrollment (n=20).
- Revision ACL Reconstruction Group: Athletes who had undergone at least two ACL surgeries including revision, with rehabilitation completed at least 6 months prior to enrollment (n=20).

SUMMARY:
This study investigated how anterior cruciate ligament (ACL) injuries affect not only the knee joint but also brain activity, reaction speed, and psychological readiness to return to sports. A total of 60 male athletes, aged 18 to 30 years, were evaluated in three groups: healthy athletes, athletes who had undergone primary ACL reconstruction, and athletes who had undergone revision ACL reconstruction.

The study measured brain activity with electroencephalography (EEG), reaction time with a computer-based test, and psychological status with standardized questionnaires. The findings showed that athletes with revision ACL surgery had more difficulties in attention control, slower reaction times, and greater psychological barriers compared to the other groups.

These results suggest that ACL injuries and surgeries may influence not only physical recovery but also brain function and psychological readiness. The study highlights the importance of considering neuromuscular, cognitive, and emotional aspects when planning rehabilitation and return-to-sport decisions.

ELIGIBILITY:
Inclusion Criteria:

Male athletes

Age between 18 and 30 years

Regular participation in amateur or professional sports

Completion of ACL rehabilitation (for surgical groups) at least 6 months before enrollment

Ability to undergo EEG and reaction time testing

Provision of signed informed consent

Exclusion Criteria:

History of neurological or psychiatric conditions (e.g., epilepsy, ADHD, depression)

Additional lower extremity injuries or orthopedic surgeries

Metal implants or scalp conditions incompatible with EEG

Uncorrected visual or auditory deficits

Systemic illnesses (e.g., diabetes, multiple sclerosis, neuropathy)

Use of psychoactive medication

Any cognitive or physical limitation interfering with testing procedures

Female participants (to avoid hormonal confounding effects on EEG recordings)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of 60 male athletes aged 18 to 30 years. Participants were divided into three groups: healthy controls with no history of knee injury, athletes with primary ACL reconstruction, and athletes with revision ACL reconstruction. All were actively engaged in regular sports participation and had completed ACL rehabilitation at least 6 months prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Frontal EEG Theta/Beta Ratio | Single assessment on the study day (June-July 2025)
  Cortical activity measured at F3 and F4 electrode sites using EEG (Nexus-10 system, Mind Media, Netherlands). Theta (4-8 Hz) and beta (13-21 Hz) power spectral densities were calculated and the ratio (theta/beta) was used as an indicator of attentional control. Higher ratios indicate reduced attention and cognitive efficiency.

SECONDARY OUTCOMES:
Visual Reaction Time (ms) | Single assessment on the study day (June-July 2025)
  Computer-based visual response task; mean reaction time (ms) computed across 5 valid trials after practice. Longer times indicate lower sensorimotor efficiency.
Kinesiophobia (TSK-11 total score) | Single assessment on the study day (June-July 2025)
  Tampa Scale of Kinesiophobia-11; 11 items, 1-4 Likert; total score 11-44. Higher scores indicate greater fear of movement/reinjury.
Psychological Readiness to Return to Sport (ACL-RSI total score) | Single assessment on the study day (June-July 2025)
  ACL-RSI questionnaire; 12 items scored 0-100; total reported as mean (0-100). Higher scores indicate greater psychological readiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset is small, contains sensitive neurophysiological and psychological information, and was collected under conditions that limit external data access. Data may be available in aggregated form upon reasonable request to the corresponding author.

REFERENCES:
- [Derived] Kaya HB, Karaduman ZO, Akpinar S, Arican M, Saglam S, Aksit S, Koc M, Uludag V. Neuromusculoskeletal alterations after ACL reconstruction: a cross-sectional study of cortical activity, motor response, and psychological readiness. BMC Sports Sci Med Rehabil. 2025 Nov 29. doi: 10.1186/s13102-025-01450-6. Online ahead of print. PMID 41318585